CLINICAL TRIAL: NCT02936635
Title: A Phase 3, Open-Label Extension Study of Tirasemtiv for Patients With Amyotrophic Lateral Sclerosis (ALS) Who Completed VITALITY-ALS (CY 4031)
Brief Title: A Study for Patients Who Completed VITALITY-ALS (CY 4031)
Acronym: VIGOR-ALS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CY 4033; 2016-002629-13 (EudraCT Number)
Record Dates: First submitted 2016-10-12; First posted 2016-10-18 (Estimated); Results first posted 2021-05-12 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Amyotrophic Lateral Sclerosis; ALS; tirasemtiv
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — CK-2017357

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delayed Start Treatment (Experimental): The Delayed Start Treatment group consisted of patients who received placebo in CY 4031 and tirasemtiv in CY 4033.
  Interventions: Drug: tirasemtiv
- Early Start Treatment (Experimental): The Early Start Treatment group consisted of patients who received tirasemtiv in both CY 4031 and CY 4033.
  Interventions: Drug: tirasemtiv

INTERVENTIONS:
Drug: tirasemtiv — Oral
  Other Names: CK-2017357

SUMMARY:
The purpose of this study is to assess the long-term safety and tolerability of tirasemtiv in patients with ALS who had completed the double-blind placebo-controlled study of tirasemtiv in ALS (CY 4031).

DETAILED DESCRIPTION:
Enrolled participants will begin dosing of tirasemtiv 125 mg twice daily (250 mg/day) for a period of 4 weeks and will titrate to their tolerated dose, the maximum dose being 250 mg twice daily (500 mg/day). This study will also compare the clinical course of patients who completed treatment with tirasemtiv in CY 4031 with those who completed treatment with placebo in CY 4031 during continued treatment of both groups with tirasemtiv during CY 4033, compare the clinical course of patients who completed treatment with tirasemtiv in CY 4031 during that study with their clinical course during continued treatment with tirasemtiv during CY 4033, and compare the clinical course of patients who completed treatment with placebo in CY 4031 during that study with their clinical course during treatment with tirasemtiv during CY 4033.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and willing to sign an Informed Consent Form (ICF). If verbal consent is given, a Legal Designee of the patient must sign the ICF form
* Completed participation on study drug and the Follow-Up Visit in the CY 4031 study
* Male patients, who have not had a vasectomy AND confirmed zero sperm count, must agree for the duration of their participation in the study to either:

  * Use a condom during sexual intercourse with female partners who are of childbearing potential AND to have female partners use a highly effective means of contraception OR
  * Abstain from sexual intercourse during participation in the study
* Female patients who are not post-menopausal (≥ 1 year) or sterilized, must:

  * Not be breastfeeding
  * Have a negative pregnancy test
  * Have no intention to become pregnant during participation in the study AND
  * Practice sexual abstinence, defined as refraining from intercourse during the duration of the study OR if male partners are not vasectomized with a confirmed zero sperm count, require use of a condom AND use of a highly effective contraceptive measure

Exclusion Criteria:

* Has a diaphragm pacing system (DPS) at study entry or anticipate DPS placement during the course of the study
* Has taken an investigational study drug (other than tirasemtiv) prior to dosing, within 30 days or five half-lives of the prior agent, whichever is greater
* Use of tizanidine and theophylline-containing medications during study participation
* Participation or planning to participate in any form of stem cell therapy for the treatment of ALS or another investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Cytokinetics, Study Director — Cytokinetics, Inc.
Locations (67):
- United States (41):
  - St. Joseph's Hospital and Medical Center - Barrow Neurology Clinics, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Irvine, Orange, California
  - UC Davis Medical Center, Sacramento, California
  - Forbes Norris MDA/ALS Research Center, San Francisco, California
  - Stanford Hospital and Clinics, Stanford, California
  - University of Colorado Hospital Anschutz Outpatient Pavilion, Aurora, Colorado
  - Hospital for Special Care, New Britain, Connecticut
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - University of Miami, Miller School of Medicine, Miami, Florida
  - Carol & Frank Morsani Center for Advanced Health Care - University of South Florida, Tampa, Florida
  - The Emory Clinic, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - University of Massachusetts Memorial Medical Center/University of Massachusetts Medical School, Worcester, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - St. Louis University, Department of Neurology & Psychiatry, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hospital for Special Surgery, New York, New York
  - Neurological Institute, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Neurosciences Institute, Neurology - Charlotte, Charlotte, North Carolina
  - Duke Neurological Disorders Clinic, Durham, North Carolina
  - Department of Neurology, Wake Forest School of Medicine, Winston-Salem, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Providence Brain and Spine Inst. ALS Center, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center - Clinical Research Center, Nashville, Tennessee
  - Texas Neurology, PA, Dallas, Texas
  - UTHSCSA - First Outpatient Research Unit, San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - West Virginia University Hospitals, Morgantown, West Virginia
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin
- UZ Leuven, Leuven, Vlaams Brabant, Belgium
- Canada (10):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Stan Cassidy Centre for Rehabilitation, Fredericton, New Brunswick
  - QE II Health Sciences, Nova Scotia Health Authority, Halifax, Nova Scotia
  - McMaster University Medical Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - Hopital Notre-Dame/CHUM, Montreal, Quebec
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
  - CHU de Quebec - Univerite' Laval, Québec, Quebec
- France (4):
  - Hopital Dupuytren, service de neurologie, Limoges
  - Hopital Gui de chauliac, Montpellier
  - CHU de Nice - Hopital Pasteur 2, Nice
  - Hopital Bretonneau, Tours
- Germany (3):
  - University of Ulm, Department of Neurology, Ulm, Baden-Wurttemberg
  - Hannover Medical School, Department of Neurology, Hanover, Lower Saxony
  - Charite Campus Virchow-Klinikum, Department of Neurology, Berlin
- Clinical Research Centre Beaumont Hospital, Dublin, Ireland
- Italy (3):
  - IRCCS Istituto Auxologico Italiano - U.O. Neurologia, Milan, Lombardy
  - Centro Clinico NEMO - Fondazione Serena Onlus, ASST Grande Ospedale Metropolitano Niguarda, Ospedale Niguarda, Milan, Lombardy
  - Dipartimento di Neuroscienze "Rita Levi Moltalcini" A.O.U. Citta della Salute e della Scienza di Torino P.O. "Molinette", Turin, Piedmont
- University Medical Center Utrecht, Utrecht, Netherlands
- Hospital Santa Maria - Centro Hospitalar Lisboa Norte, Lisbon, Portugal
- Hospital San Rafael, Madrid, Spain
- King's College Hospital NHS Foundation Trust, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with ALS were enrolled at 69 sites in Belgium, Canada, France, Germany, Ireland, Italy, Netherlands, Portugal, Spain, the United Kingdom, and the United States. The study was conducted from 17 October 2016 (date first patient enrolled) through 26 October 2018 (date of last patient contact).
Pre-assignment Details: Eligible patients completed participation in Study CY 4031 on study drug and had completed the scheduled follow-up visit for that study.
Period: Overall Study
Arm/Group | Delayed Start Treatment | Early Start Treatment
Started | 115 | 165
Completed | 0 | 0
Not Completed | 115 | 165
Not completed — Adverse Event | 43 | 25
Not completed — Progressive Disease | 10 | 18
Not completed — Sponsor Discretion | 10 | 16
Not completed — Death | 9 | 15
Not completed — Withdrawal by Subject | 8 | 15
Not completed — Physician Decision | 2 | 9
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Lack of effect/Entry into other study | 31 | 65

BASELINE CHARACTERISTICS:
Population: The data provided are for the Efficacy Analysis Set, which consisted of patients who completed CY 4031, were enrolled in CY 4033, received at least 1 dose of tirasemtiv, and had at least one post-baseline efficacy outcome assessment during CY 4033.
Groups:
- Total: Total of all reporting groups
Arm/Group | Delayed Start Treatment | Early Start Treatment | Total
Number analyzed (Participants) | 111 | 162 | 273
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (10.07) | 57.7 (9.13) | 56.9 (9.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 46 | 81
  Male | 76 | 116 | 192
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 105 | 158 | 263
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Time since ALS symptom onset at screening in parent study [Mean (Standard Deviation); unit: months] | 23.60 (17.078) | 19.15 (11.041) | 20.96 (13.961)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: The number of participants with adverse events was used as the measure for the long-term safety and tolerability of tirasemtiv.
Time Frame: From the first dose of tirasemtiv through 28 days after the last dose
Population: The data are presented for the Safety Analysis Set, which consisted of all patients who enrolled and received at least 1 dose of tirasemtiv in Study CY 4033.
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed Start Treatment | Early Start Treatment
Number analyzed (Participants) | 115 | 165
Participants | 112 | 157

2. Secondary Outcome: Change From CY 4031 Baseline in Percent Predicted Slow Vital Capacity to Week 24 in CY 4033
Description: Slow vital capacity (SVC) was measured using a spirometer (in units of liters). Following 3 to 5 breaths at rest, patients were instructed to take as deep an inspiration as possible followed by a maximum exhalation (blowing out all the air in their lungs). Values obtained were converted to percent predicted values (ie, the test result as a percent of predicted values for patients of similar demographic and baseline characteristics [eg, height, age, sex]).
Time Frame: baseline and 24 weeks
Population: The analysis population includes patients who received at least 1 dose of tirasemtiv and had slow vital capacity results at Week 24.
Measure: Least Squares Mean (Standard Error); unit: change in % predicted SVC
Arm/Group | Delayed Start Treatment | Early Start Treatment
Number analyzed (Participants) | 48 | 94
change in % predicted SVC | -28.79 (2.845) | -32.69 (2.285)
Statistical Analysis 1: Comparison: Delayed Start Treatment vs Early Start Treatment; Test type: Superiority; p = 0.2821, Mixed Models Analysis; Mean Difference (Final Values) = -3.9, 95% CI 2-sided [-11.035 to 3.23], Standard Error of Mean 3.619

3. Secondary Outcome: Change From CY 4031 Baseline in Percent Predicted Slow Vital Capacity to Week 48 in CY 4033
Description: Slow vital capacity was measured using a spirometer (in units of liters). Following 3 to 5 breaths at rest, patients were instructed to take as deep an inspiration as possible followed by a maximum exhalation (blowing out all the air in their lungs). Values obtained were converted to percent predicted values (ie, the test result as a percent of predicted values for patients of similar demographic and baseline characteristics [eg, height, age, sex]).
Time Frame: baseline and 48 weeks
Population: The analysis population includes patients who received at least 1 dose of tirasemtiv and had slow vital capacity results at Week 48.
Measure: Least Squares Mean (Standard Error); unit: percent predicted slow vital capacity
Arm/Group | Delayed Start Treatment | Early Start Treatment
Number analyzed (Participants) | 28 | 45
percent predicted slow vital capacity | -35.55 (3.332) | -40.87 (2.667)
Statistical Analysis 1: Comparison: Delayed Start Treatment vs Early Start Treatment; Test type: Superiority; p = 0.2118, Mixed Models Analysis; Median Difference (Final Values) = -5.32, 95% CI 2-sided [-13.711 to 3.067], Standard Error of Mean 4.242

4. Secondary Outcome: Change From CY 4031 Baseline in ALS Functional Rating Scale - Revised (ALSFRS-R) Total Score at Week 24
Description: The ALSFRS-R is used to measure the progression and severity of disability in patients with ALS. The ALSFRS-R consists of 12 questions, assessing a patient's capability and independence in functional activities relevant to ALS, categorized in the following 4 domains: gross motor tasks, fine motor tasks, bulbar functions, and respiratory function. Each question is scored from 0 (indicating incapable or dependent) to 4 (normal). The total score ranges from 0 to 48, with higher scores reflecting more normal function and lower scores reflecting more impaired function. Comparing postbaseline to baseline assessments, a negative value indicates a worsening in function.
Time Frame: baseline and 24 weeks
Population: The analysis population includes patients who received at least 1 dose of tirasemtiv and had an ALSFRS-R total score at Week 24.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Delayed Start Treatment | Early Start Treatment
Number analyzed (Participants) | 75 | 120
scores on a scale | -13.78 (0.934) | -14.35 (0.767)
Statistical Analysis 1: Comparison: Delayed Start Treatment vs Early Start Treatment; Test type: Superiority; p = 0.6354, Mixed Models Analysis; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-2.946 to 1.801], Standard Error of Mean 1.205

5. Secondary Outcome: Change From CY 4031 Baseline in ALSFRS-R Total Score at Week 48
Description: as for outcome 4
Time Frame: baseline and 48 weeks
Population: The analysis population includes patients who received at least 1 dose of tirasemtiv and had an ALSFRS-R total score at Week 48.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Delayed Start Treatment | Early Start Treatment
Number analyzed (Participants) | 38 | 62
scores on a scale | -17.61 (1.171) | -17.82 (0.956)
Statistical Analysis 1: Comparison: Delayed Start Treatment vs Early Start Treatment; Test type: Superiority; p = 0.8887, Mixed Models Analysis; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-3.186 to 2.763], Standard Error of Mean 1.509

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the first administration of tirasemtiv through 28 days after the last dose of tirasemtiv.
Description: An AE was treatment-emergent if it started after initiation of study drug dosing in CY 4033 or was present at initiation of study drug dosing in CY 4033 and subsequently worsened in severity.
Arm/Group | Delayed Start Treatment | Early Start Treatment
All-Cause Mortality (participants affected / at risk) | 21/115 | 28/165
Serious Adverse Events (participants affected / at risk) | 32/115 | 53/165
Other Adverse Events (participants affected / at risk) | 111/115 | 155/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delayed Start Treatment (N=115) | Early Start Treatment (N=165)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (8)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 9 (9)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Amyotrophic lateral sclerosis (Nervous system disorders) | 4 (4) | 13 (14)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Euthanasia (General disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (3) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delayed Start Treatment (N=115) | Early Start Treatment (N=165)
Dizziness (Nervous system disorders) | 49 (73) | 44 (63)
Somnolence (Nervous system disorders) | 28 (33) | 27 (35)
Headache (Nervous system disorders) | 8 (8) | 14 (17)
Dysarthria (Nervous system disorders) | 7 (9) | 6 (7)
Constipation (Gastrointestinal disorders) | 20 (26) | 33 (38)
Nausea (Gastrointestinal disorders) | 19 (21) | 22 (28)
Dysphagia (Gastrointestinal disorders) | 12 (13) | 9 (9)
Salivary hypersecretion (Gastrointestinal disorders) | 8 (9) | 10 (12)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 12 (14)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 4 (4)
Fatigue (General disorders) | 42 (58) | 51 (65)
Asthenia (General disorders) | 14 (17) | 8 (11)
Oedema peripheral (General disorders) | 6 (8) | 6 (6)
Feeling abnormal (General disorders) | 6 (7) | 4 (6)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 16 (25) | 33 (45)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 18 (20) | 10 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6) | 9 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 7 (7)
Fall (Injury, poisoning and procedural complications) | 22 (44) | 23 (45)
Contusion (Injury, poisoning and procedural complications) | 11 (17) | 13 (20)
Skin abrasion (Injury, poisoning and procedural complications) | 9 (11) | 4 (9)
Post-traumatic pain (Injury, poisoning and procedural complications) | 6 (9) | 4 (4)
Anxiety (Psychiatric disorders) | 16 (19) | 12 (13)
Insomnia (Psychiatric disorders) | 16 (16) | 14 (16)
Depression (Psychiatric disorders) | 16 (19) | 10 (11)
Confusional state (Psychiatric disorders) | 8 (10) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (17) | 16 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 7 (9)
Choking (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 4 (5)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
Nasopharyngitis (Infections and infestations) | 8 (10) | 18 (22)
Urinary tract infection (Infections and infestations) | 5 (6) | 10 (10)
Weight decreased (Investigations) | 13 (15) | 9 (9)
Decreased appetite (Metabolism and nutrition disorders) | 16 (19) | 13 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-07-13): https://cdn.clinicaltrials.gov/large-docs/35/NCT02936635/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/35/NCT02936635/SAP_001.pdf